CLINICAL TRIAL: NCT06721455
Title: Mathematical Modeling of Salvaged Red Blood Cells-based Blood Management Strategy and Their Hemolytic Risk in Pediatric Cardiac Surgery
Brief Title: Modeling Blood Management and Hemolytic Risk in Pediatric Heart Surgery
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, MD, Boston Children's Hospital
Other Study IDs: IRB-P00049726
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Heart Surgery; Blood Transfusion; Hemolysis
MeSH Terms: conditions — Hemolysis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Discarded blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children having heart surgery: Children under 18 years of age having heart surgery with cardio-pulmonary bypass at Boston Children's Hospital
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Discarded blood samples will be taken from routine clinical labs drawn during and after heart surgery.

SUMMARY:
This study aims to learn more about blood management in children undergoing heart surgery, such as the right amounts, and the best blood products, to administer. It also aims to develop a mathematical model that may help researchers better predict and treat patients who need blood transfusions during heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients under 18 years of age undergoing cardiac surgery with clear prime on cardio-pulmonary bypass (CPB) at Boston Children's Hospital (BCH).

Exclusion Criteria:

* patients with known hemolytic disorders, patients on nitric oxide preoperatively, and patients found to have abnormal coagulation on routine preoperative assessment. Patients receiving heparin, American Society of Anesthesia (ASA) status, apixaban, warfarin, or bivalirudin held appropriately (i.e. for elective surgery) will not be excluded

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients under 18 years of age undergoing cardiac surgery with clear prime on cardio-pulmonary bypass (CPB) at Boston Children's Hospital (BCH).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative hemolysis during pediatric cardiac cardio-pulmonary bypass (CPB) cases as assessed using the plasma free hemoglobin assessment | 1 day (during cardio-pulmonary bypass)

SECONDARY OUTCOMES:
In vitro salvaged red blood cells (RBCs) co-incubation with patients' plasma for hemolysis assessment compared to patients' baseline RBCs | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No